CLINICAL TRIAL: NCT01670760
Title: 3M(TM)SpotOn(TM) Temperature Monitoring System Thermometry Trial
Brief Title: Zero Heat Flux Thermometry System Comparison Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-DTT-BS-01
Record Dates: First submitted 2012-08-16; First posted 2012-08-22 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Body Temperature; Thermosensing; Temperature
Keywords: Deep Tissue Temperature; Zero Heat Flux Thermometry; Thermometry; Core Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zero-Heat-Flux (Experimental): This is a single arm study. All patients will have deep tissue temperature monitored from the nasopharyngeal and lateral forehead sites simultaneously.
  Interventions: Device: Zero-heat-flux thermometry

INTERVENTIONS:
Device: Zero-heat-flux thermometry — The zero-heat-flux thermometer will be placed on the subject's lateral forehead for the duration of the surgery to measure deep tissue temperature.
  Other Names: 3M(TM) SpotOn(TM) temperature monitoring system

SUMMARY:
Nasopharyngeal and deep tissue temperatures will be measured simultaneously during surgery and compared for agreement. The hypothesis of this trial is that deep tissue temperature as measured by zero-heat-flux thermometry will agree with nasopharyngeal temperatures during surgery.

DETAILED DESCRIPTION:
The core temperature of the body normally decreases in response to anesthesia. Deep tissue temperature can be used to estimate of body core temperature. Deep tissue temperature of the forehead will be measured using a new technology known as zero-heat-flux thermometry. The usual way to measure internal body temperature is within the nasal cavity (nasopharyngeal temperature). Nasopharyngeal and deep tissue temperatures will be measured simultaneously during surgery and compared for agreement. The hypothesis of this trial is that deep tissue temperature as measured by zero-heat-flux thermometry will agree with nasopharyngeal temperatures during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 17 years old
* patients undergoing surgery during which core temperature is estimated
* Willing to participate in trial
* Able to provide consent
* Adequate forehead surface area available for probe attachment
* Urology, orthopedic, or general abdominal surgery

Exclusion Criteria:

* Skin lesions at thermometer target site
* Infectious disease
* Bleeding disorder
* Prone intraoperative positioning anticipated
* Head and neck procedures
* Cardiothoracic procedures
* Tonsillectomy, cosmetic, or other brief surgical or nonsurgical procedures

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Davis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburg of the University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Langham GE, Maheshwari A, Contrera K, You J, Mascha E, Sessler DI. Noninvasive temperature monitoring in postanesthesia care units. Anesthesiology. 2009 Jul;111(1):90-6. doi: 10.1097/ALN.0b013e3181a864ca. PMID 19512860
- [Background] Teunissen LP, Klewer J, de Haan A, de Koning JJ, Daanen HA. Non-invasive continuous core temperature measurement by zero heat flux. Physiol Meas. 2011 May;32(5):559-70. doi: 10.1088/0967-3334/32/5/005. Epub 2011 Mar 28. PMID 21444968
- [Background] Fox RH, Solman AJ. A new technique for monitoring the deep body temperature in man from the intact skin surface. J Physiol. 1971 Jan;212(2):8P-10P. No abstract available. PMID 5548025
- [Background] Togwa T, Nemoto T, Yamazaki T, Kobayashi T. A modified internal temperature measurement device. Med Biol Eng. 1976 May;14(3):361-4. doi: 10.1007/BF02478138. No abstract available. PMID 940402
- [Background] Matsukawa T, Sessler DI, Ozaki M, Hanagata K, Iwashita H, Kumazawa T. Comparison of distal oesophageal temperature with "deep" and tracheal temperatures. Can J Anaesth. 1997 Apr;44(4):433-8. doi: 10.1007/BF03014466. PMID 9104528
- [Background] Harioka T, Matsukawa T, Ozaki M, Nomura K, Sone T, Kakuyama M, Toda H. "Deep-forehead" temperature correlates well with blood temperature. Can J Anaesth. 2000 Oct;47(10):980-3. doi: 10.1007/BF03024869. PMID 11032273
- [Background] Yamakage M, Namiki A. Deep temperature monitoring using a zero-heat-flow method. J Anesth. 2003;17(2):108-15. doi: 10.1007/s005400300026. No abstract available. PMID 12903922
- [Background] Jost U, Hanf K, Kohler CO, Just OH. [A new method for the transcutaneous measurement of deep body temperature during anaesthesia and intensive care (author's transl)]. Prakt Anaesth. 1978 Apr;13(2):144-9. German. PMID 652707
- [Background] Esamai F, Mining S, Forsberg P, Lewis DH. A comparison of brain, core and skin temperature in children with complicated and uncomplicated malaria. J Trop Pediatr. 2001 Jun;47(3):170-5. doi: 10.1093/tropej/47.3.170. PMID 11419682
- [Background] Akata T, Setoguchi H, Shirozu K, Yoshino J. Reliability of temperatures measured at standard monitoring sites as an index of brain temperature during deep hypothermic cardiopulmonary bypass conducted for thoracic aortic reconstruction. J Thorac Cardiovasc Surg. 2007 Jun;133(6):1559-65. doi: 10.1016/j.jtcvs.2006.11.031. PMID 17532957
- [Background] Yamakage M, Iwasaki S, Namiki A. Evaluation of a newly developed monitor of deep body temperature. J Anesth. 2002;16(4):354-7. doi: 10.1007/s005400200056. No abstract available. PMID 14517632

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zero-Heat-Flux
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zero-Heat-Flux
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Body Temperature Difference in Degrees Celsius
Description: Body temperature difference as defined by Agreement (bias - Zero heat flux thermometry minus nasopharyngeal) between simultaneously-acquired nasopharyngeal and forehead deep tissue temperatures as assessed by Bland and Altman repeated measures technique.
Time Frame: Every 5 to 10 minutes, or as clinically indicated, for the duration of the surgery from the time of incision to the time of closure. The average duration of surgery was 57 minutes.
Measure: Least Squares Mean (Standard Error); unit: Degrees Celsius
Units Other Than Participants: Observation
Arm/Group | Zero-Heat-Flux
Number analyzed (Participants) | 20
Number analyzed (Observation) | 247
Degrees Celsius | -0.28 (0.027)
Statistical Analysis 1: Comparison: Zero-Heat-Flux; Test type: Superiority or Other; p = 0.69, ANOVA; Mean Difference (Final Values) = 0.69

ADVERSE EVENTS:
Time Frame: For the duration of the surgery from the time of incision to the time of closure. The average duration of surgery was 57 minutes.
Arm/Group | Zero-Heat-Flux
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 11/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zero-Heat-Flux (N=20)
Redness at attachment site (Skin and subcutaneous tissue disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No